CLINICAL TRIAL: NCT05330078
Title: Examining the Therapeutic Potential of Botulinum Toxin Type A in the Treatment of Keloids
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Arisa Ortiz, Principal investigator, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201088
Record Dates: First submitted 2022-03-16; First posted 2022-04-15 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Keloid
MeSH Terms: conditions — Keloid | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a single center, randomized, single-masked, prospective experimental study. Half the keloid tissue will be treated with Botulinum toxin type A while the other half will be treated with a vehicle control (saline) of matching number of injections and volume. All treated keloids will serve as their own internal control. The treatment and control sides of the keloid will clearly be documented in the patient's chart and source documents to allow the study physician to track treatment vs vehicle control portions of the keloid.
Who Masked: Participant, Outcomes Assessor
Masking Description: Keloid treatment will be randomized. Participants will not be informed of which side will be treated with botulinum toxin type A vs vehicle control (saline).
  Blinded physician evaluators will not have access to information regarding keloid treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Keloid treatment with botulinum toxin type A (Experimental): Participants will receive Botulinum toxin type A 5 units / cm3 with injections of 0.2mL spaced evenly 1cm apart within the treatment area (half of the keloid). Each treatment will consist of a maximum of 2 mL (10 injection sites, 50 unit total) of the study drug. Patients will undergo 3 treatments, 6 weeks apart.
  Interventions: Drug: Botulinum toxin type A
- Keloid treatment with vehicle control (saline) (Placebo Comparator): Participants will receive saline injections of 0.2mL spaced evenly 1cm apart within the placebo area (half of the keloid). Each treatment will consist of a maximum of 2 mL (10 injection sites) of the vehicle control (saline). Patients will undergo 3 treatments, 6 weeks apart.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Botulinum toxin type A — Participants will receive Botulinum toxin type A 5 units / cm3 with injections of 0.2mL spaced evenly 1cm apart within the treatment area (half of the keloid). Each treatment will consist of a maximum of 2 mL (10 injection sites, 50 unit total) of the study drug. Patients will undergo 3 treatments, 6 weeks apart.
  Arms: Keloid treatment with botulinum toxin type A
Drug: Vehicle — Participants will receive saline injections of 0.2mL spaced evenly 1cm apart within the placebo area (half of the keloid). Each treatment will consist of a maximum of 2 mL (10 injection sites) of the vehicle control (saline). Patients will undergo 3 treatments, 6 weeks apart.
  Other Names: vehicle control (saline)
  Arms: Keloid treatment with vehicle control (saline)

SUMMARY:
Keloids are a common form of hypertrophic scars that by definition last beyond 6 months and grow beyond the site of initial injury. Keloids are a common complaint from patients in dermatology and cause significant functional impairment due to cosmetic disfigurement, itching and pain. Current treatment modalities include intralesional corticosteroids, chemotherapeutic agents and laser therapy. Initial reports have demonstrated that Botulinum toxin type A may be a viable treatment option for keloids that can reduce keloid size and reduce associated symptoms while having fewer side effects when compared to intralesional corticosteroid injection, which can cause unnatural blood vessel growth or skin thinning. To date, no study has carefully examined the efficacy of Botulinum toxin type A in treating keloids or its mechanistic effects on keloid biology. Our aim in this study is to pursue a rigorous, randomized control trial to assess the potential use Botulinum toxin type A to treat keloids. Efficacy will be objectively be mentioned by change in keloid size after treatment, along with subjective measures of patient satisfaction and symptoms, and finally physician rated scores. Also, samples from three patients will be analyzed in the laboratory setting to determine the underlying molecular mechanism behind the effects of Botulinum toxin type A on keloid biology.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 80
2. History of keloid scar for at least 12 months
3. Absence of keloid treatment for past 12 months
4. Participant must have a keloid scar of at least 4cm in length.
5. Participants who score at least 8 or higher on the Vancouver Scar Scale
6. Subjects who score 5 (neither satisfied nor dissatisfied) to 10 (maximally dissatisfied) on the patient subjective score of dissatisfaction with keloid.
7. Participants must be in stable health, as confirmed by medical history, per investigator judgment
8. Participants must be able to read, sign, and understand the informed consent
9. Participants must be willing to avoid any other treatments to the keloid that will be treated including corticosteroid injections, surgical excision, chemotherapeutic injection, lasers, light-based therapy, radiation therapy, cryotherapy, or pressure therapy, during the study period.

Exclusion Criteria:

1. Pregnant women
2. Keloids on face, neck or scalp
3. History of hypersensitivity to botulinum toxin
4. Ongoing or planned treatment with chemotherapy, radiation, isotretinoin, cytokine-based immunotherapies
5. Any planned surgery during study period
6. Known diagnosis of insulin dependent diabetes mellitus
7. Patients being treating with dupilumab for any indication
8. Patients taking aminoglycoside antibiotics
9. Patients with pre-existing neuromuscular disorders
10. Patients with infection around potential injection sites

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Keloid volume | Measurements obtained at 0 and 24 weeks.
  Keloid volume will be measured using the high resolution 3D imaging system (Cherry Imaging platform)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Publication will be submitted in a peer reviewed journal.

REFERENCES:
- [Background] Bi M, Sun P, Li D, Dong Z, Chen Z. Intralesional Injection of Botulinum Toxin Type A Compared with Intralesional Injection of Corticosteroid for the Treatment of Hypertrophic Scar and Keloid: A Systematic Review and Meta-Analysis. Med Sci Monit. 2019 Apr 22;25:2950-2958. doi: 10.12659/MSM.916305. PMID 31006769
- [Background] Cocco A, Albanese A. Recent developments in clinical trials of botulinum neurotoxins. Toxicon. 2018 Jun 1;147:77-83. doi: 10.1016/j.toxicon.2017.08.014. Epub 2017 Aug 14. PMID 28818530
- [Background] Shaarawy E, Hegazy RA, Abdel Hay RM. Intralesional botulinum toxin type A equally effective and better tolerated than intralesional steroid in the treatment of keloids: a randomized controlled trial. J Cosmet Dermatol. 2015 Jun;14(2):161-6. doi: 10.1111/jocd.12134. Epub 2015 Mar 24. PMID 25810045